CLINICAL TRIAL: NCT00397202
Title: FLOW-Finding Lasting Options for Women: A Prospective, Randomized, Multicenter Trial Comparing Tampons to a Menstrual Cup
Brief Title: FLOW-Finding Lasting Options for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Research System-College of Family Physicians of Canada (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H06-70478
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Menstruation
Keywords: Menstruation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The DivaCupTM (Active Comparator)
  Interventions: Device: Diva Cup TM

INTERVENTIONS:
Device: Diva Cup TM — See Detailed Description.

SUMMARY:
1. Purpose: To compare the use of the menstrual cup "The DivaCupTM " to a menstrual strategy using tampons as the primary method of menstrual flow management using indicators of user-satisfaction, urinary tract infection, vaginal irritation, cost and waste.
2. Hypothesis: The "The DivaCupTM" will have similar rates of user-satisfaction, urinary tract infection, and vaginal irritation as a menstrual strategy using tampons as the primary method of menstrual flow management but will likely be more reasonable in terms of cost and will generate less waste.

DETAILED DESCRIPTION:
Method:

Prospective study of 100 women from family practice offices in Vancouver, Victoria and Prince George who currently use tampons to manage menstrual flow. After an information session and consent, subjects will be randomized to tampon use or Diva Cup use and record their experience on a diary for 3 months. Women who attend the information session and who do not enrol, or those who drop out will be asked their reasons for discontinuing, and their pre-study questionnaire will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 19 and 40 who have menstrual flow most months and who currently self-identify as using tampons as their primary method of menstrual management

Exclusion Criteria:

* Have a sensitivity or allergy to silicone
* Have an active vaginal or urogenital infection
* Are pregnant, or who have plans to become pregnant before spring 2007 (end of study data collection)
* Have used systemic antimicrobials within the previous 14 days
* Are unable to understand the nature and purpose of the study
* Are unable to understand and express themselves in written and spoken English

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction with menstrual strategy.

SECONDARY OUTCOMES:
Diagnosed UTI
Diagnosed vaginitis
Vaginal irritation
Waste
Cost

CONTACTS AND LOCATIONS:
Overall Officials: Konia Trouton, MD, Principal Investigator — University of British Columbia
Locations (1):
- Private family physician offices, Victoria, Vancouver, Prince George, British Columbia, Canada

REFERENCES:
- [Derived] Howard C, Rose CL, Trouton K, Stamm H, Marentette D, Kirkpatrick N, Karalic S, Fernandez R, Paget J. FLOW (finding lasting options for women): multicentre randomized controlled trial comparing tampons with menstrual cups. Can Fam Physician. 2011 Jun;57(6):e208-15. PMID 21673197